CLINICAL TRIAL: NCT05418023
Title: Validation of a Salivary miRNA Diagnostic Test for Autism Spectrum Disorder
Brief Title: Validation of a Salivary miRNA Diagnostic Test for ASD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Quadrant Biosciences Inc. (Industry)
Collaborators: University of California, Irvine (Other); Holland Bloorview Kids Rehabilitation Hospital (Other); Children's Hospital of Philadelphia (Other); MetroHealth Medical Center (Other); University of Rochester (Other); Nationwide Children's Hospital (Other); Children's Hospital Medical Center, Cincinnati (Other); University of Pittsburgh (Other); University of Massachusetts, Worcester (Other); Children's Hospital Los Angeles (Other); Prisma Health-Upstate (Other); University of Virginia (Other); State University of New York - Upstate Medical University (Other); Rush University (Other); Seattle Children's Hospital (Other); Drexel University (Other); Emory University (Other)
Responsible Party: Sponsor
Other Study IDs: 20214744
Record Dates: First submitted 2022-01-06; First posted 2022-06-14 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Autism Spectrum Disorder; Developmental Delay
Keywords: Autism Spectrum Disorder; ASD; Saliva; Biomarkers
MeSH Terms: conditions — Autism Spectrum Disorder; Learning Disabilities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Autism Spectrum Disorder (ASD)
  Interventions: Other: Salivary Collection; Other: Adaptive Assessment; Other: Medical and Demographic questionnaire; Other: Autism Assessment; Other: Intellectual Development Assessment
- Non-ASD
  Interventions: Other: Salivary Collection; Other: Adaptive Assessment; Other: Medical and Demographic questionnaire; Other: Autism Assessment; Other: Intellectual Development Assessment

INTERVENTIONS:
Other: Salivary Collection — Collection of saliva via swab for miRNA processing
Other: Adaptive Assessment — Includes Vineland Adaptive Behavior Scale or equivalent
Other: Medical and Demographic questionnaire — Survey that collects basic medical and demographic information
Other: Autism Assessment — Includes Autism Diagnostic Observation Schedule (ADOS), Childhood Autism Rating Scale (CARS), Gilliam Autism Rating Scale (GARS), Autism Diagnostic Interview - Revised (ADIR) or an equivalent
Other: Intellectual Development Assessment — Includes Mullens Scales of Early Learning, Stanford Binet Intelligence Scales, Wechsler Preschool and Primary Scale of Intelligence (WPPSI), Bayley Scales of Infant Development or an equivalent

SUMMARY:
This study involves sample collection to identify biomarkers relating to Autism Spectrum Disorder(ASD) in the saliva of children who are between the ages of 18 months to 6 years and 11 months. Participants will at each timepoint have a non-invasive saliva swab collected and complete a brief demographic and medical history questionnaire as well. Children in the pediatric/provider setting who will receive a referral for an ASD diagnosis because they were determined to have a suspicion of developing ASD will be enrolled in the study. Children will also be enrolled in the specialist evaluation setting where they will receive a DSM-5 diagnosis. A subset of both enrollment cohorts will also be followed up with at a third time point in which their diagnosis will be confirmed, and information about any ongoing treatment will be gathered.

ELIGIBILITY:
Inclusion Criteria:

* 18 through 83 months old
* The study will include children "at risk" for ASD as defined by meeting one or more of the following criteria:

  * flagged positive on a developmental screening tool (see below for assessment cut off scores)
  * the child has a biological sibling with ASD
  * Significant provider concern based on parent report noted in the child's medical chart at the time of the appointment.
  * Significant parental concern

Exclusion Criteria:

* Feeding tube dependence
* Active periodontal disease
* Confounding neurological condition (i.e. cerebral palsy, epilepsy)
* Sensory impairments (i.e. blindness or deafness)
* Acute illnesses (i.e. upper respiratory infection)
* Currently on antibiotics
* Had taken antibiotics within the previous 30 days
* Wards of the state

Ages: 18 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants will be enrolled at pediatric offices, as well as specialist evaluation centers who are deemed at-risk for Autism Spectrum Disorder.
Sampling Method: Non-Probability Sample
Enrollment: 6604 (Estimated)
Dates: Start 2022-03-16 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Salivary miRNA Profile | At the time of collection (from 18 months to 6 years 11 months of age)
  Measures of miRNA abundance in saliva
DSM-5 Diagnosis | At the time of the diagnostic evaluation
  Confirmation of participants meeting or not meeting the DSM-5 Criteria for a diagnosis of Autism Spectrum Disorder

CONTACTS AND LOCATIONS:
Overall Officials: David Levitskiy, MS, Principal Investigator — Quadrant Biosciences
Locations (16):
- United States (16):
  - University of California - Irvine, Santa Ana, California
  - Marcus Autism Center/Emory University, Atlanta, Georgia
  - RUSH University, Chicago, Illinois
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - University of Rochester, Rochester, New York
  - Quadrant Biosciences, Syracuse, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - MetroHealth Medical Center, Parma, Ohio
  - Nationwide Children's Hospital, Westerville, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Drexel University, Philadelphia, Pennsylvania
  - Prisma Health-Upstate, Greenville, South Carolina
  - Texas Children's Hospital/Baylor College of Medicine, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- [Background] Hicks SD, Ignacio C, Gentile K, Middleton FA. Salivary miRNA profiles identify children with autism spectrum disorder, correlate with adaptive behavior, and implicate ASD candidate genes involved in neurodevelopment. BMC Pediatr. 2016 Apr 22;16:52. doi: 10.1186/s12887-016-0586-x. PMID 27105825
- [Background] Hicks SD, Rajan AT, Wagner KE, Barns S, Carpenter RL, Middleton FA. Validation of a Salivary RNA Test for Childhood Autism Spectrum Disorder. Front Genet. 2018 Nov 9;9:534. doi: 10.3389/fgene.2018.00534. eCollection 2018. PMID 30473705
- [Background] Hicks SD, Carpenter RL, Wagner KE, Pauley R, Barros M, Tierney-Aves C, Barns S, Greene CD, Middleton FA. Saliva MicroRNA Differentiates Children With Autism From Peers With Typical and Atypical Development. J Am Acad Child Adolesc Psychiatry. 2020 Feb;59(2):296-308. doi: 10.1016/j.jaac.2019.03.017. Epub 2019 Mar 27. PMID 30926572